CLINICAL TRIAL: NCT01823237
Title: Effect of Increasing Motor Cortex Inhibition on Task Specific Dystonia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is temporarily suspended pending additional funding to continue subject recruitment.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Cathrin Buetefisch, Associate Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB00062538; DYST (Other: Other)
Record Dates: First submitted 2013-03-19; First posted 2013-04-04 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Dystonia
Keywords: Dystonia; Transcranial Magnetic Stimulation; Rehabilitation; Plasticity
MeSH Terms: conditions — Dystonia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS (Active Comparator): rTMS condition, rTMS will be applied at 0.1-0.5 Hz frequency at a subthreshold intensity
  Interventions: Device: Transcranial Magnetic Stimulation
- rTMS sham (Placebo Comparator): Placebo condition will use a sham coil and apply a very small magnetic stimulus
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation
  Other Names: TMS

SUMMARY:
Dystonia is a disease where muscles in the affected body part are abnormally active. This may result in abnormal postures. The underlying mechanisms are not known. One proposed mechanism is located in the motor area of the brain that controls the coordination of muscles, called the motor cortex. It is well known that the motor area of one hemisphere of the brain (motor cortex) controls the movement of the opposite side of the body. When people perform tasks such as picking up an object or writing there are mechanisms in motor cortex that focus the level of activity so that they can do these tasks with a high level of precision. Focusing activity in motor cortex seems to be disturbed in people with dystonia. Transcranial magnetic stimulation (TMS) is a device that allows the non-invasive stimulation of the brain. When applied to the motor cortex it can upregulate or down regulate its activity. In the present study the investigators will conduct experiments on subjects with task specific focal hand dystonia (such as writers cramp) using TMS to decrease unwanted motor activity. The investigators will assess the effects of this intervention using objective, subjective and kinematic measures. This is a pilot study and will require further research to assess the long-term effects of repetitive TMS on task-specific focal hand dystonia.

ELIGIBILITY:
Inclusion Criteria:

* If you are treated with Botulinum toxin, the testing should be done at least 3 months after your last Botulinum toxin injections.
* Adult patients with task-specific dystonia strictly confined to one hand since the onset of symptoms
* No dystonic movements at rest
* Normal MRI scan of the brain as per clinical record
* No intake of CNS active drugs that may interfere with the study
* No contraindication for TMS
* Ability to perform the selective task
* No other neurological disease that may interfere with the study
* Ability to give informed consent

Exclusion Criteria:

* You have a history of migraines
* You have a diagnosed seizure disorder
* You take any Central Nervous System CNS active drugs, such as benzodiazepines, Lorazepam, Baclofen, SSRI's and other anti-depressants, etc. that may interfere with the response to TMS.
* You have any clips or implants in your head
* You have a pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy of TMS on task-specific focal hand dystonia | Up to 3 weeks (2 visits)
  We will assess the effects of rTMS using objective, subjective and kinematic measures. This is a pilot study and will require further research to assess the long-term effects of repetitive TMS on task-specific focal hand dystonia.

CONTACTS AND LOCATIONS:
Overall Officials: Cathrin Buetefisch, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States